CLINICAL TRIAL: NCT04254848
Title: Evaluation of Oral Stereognosis in Completely Edentulous Patient With Maxillary Tori
Brief Title: Oral Stereognosis in Completely Edentulous Patient With Maxillary Tori
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Segi University (Other)
Responsible Party: Principal Investigator, Indumathi Sivakumar, Research Supervisor and Principal investigator, Segi University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: SEGiEC/SR/FOD/2018-19/10
Record Dates: First submitted 2020-01-20; First posted 2020-02-05 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Torus Palatinus and Torus Mandibularis
Keywords: oral stereognosis; completely edentulous
MeSH Terms: conditions — Torus Palatinus and Torus Mandibularis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- completely edentulous patients with maxillary tori (Experimental): 20 completely edentulous patients with maxillary tori will be recruited for the study. The oral stereognosis will be evaluated by oral stereognostic test which employs manipulation and identification 6 different test pieces when placed in the patients mouth.
  Interventions: Other: oral stereognostic test
- completely edentulous patients without maxillary tori (Active Comparator): 20 completely edentulous patients without maxillary tori will serve as control group for the study. The oral stereognosis will be evaluated by oral stereognostic test which employs manipulation and identification 6 different test pieces when placed in the patients mouth.
  Interventions: Other: oral stereognostic test

INTERVENTIONS:
Other: oral stereognostic test — Six test pieces were selected from the 20 shapes of test pieces from National Institute of Dental Research. The test pieces comprises of 6 shaped forms which include circle, plus, square, rectangular, triangle and toroid shaped. A 2mm stainless steel wire was bent forming the test piece shape following the standard dimensions (13mm length and 2mm thickness)as described by National Institute of Dental Research to serve as the test pieces mould. Using the six test piece moulds, light cured acrylic resin test samples were fabricated. The test samples were trimmed and polished to meet the standardized measurements. A total of 240 test sample (6 samples for each patient) for 20 completely edentulous patients with maxillary tori and 20 completely edentulous patients without tori were made for the study. The test pieces were attached to dental floss to prevent any accidentally aspiration during the study.
  Other Names: oral stereognostic ability

SUMMARY:
This study aimed to evaluate the oral stereognosis in completely edentulous patients with palatal tori. Oral stereognosis is tested using different test specimens in completely edentulous patients with maxillary tori and completely edentulous patients without maxillary tori.

DETAILED DESCRIPTION:
Oral Stereognosis has been defined as appreciation of the form of objects that is explored intra-orally. In this study the oral stereognosis is determined by placing objects of various shapes in the patient's mouth and having the patient identify the correct form. Several studies has proved that oral stereognosis ability (OSA) can be used as a predictor for determining the ability of the patients with missing teeth to adapt to a new prosthesis placed in the patient's mouth.

Maxillary tori is a non-cancerous bony swelling found in palate and have high prevalence among Malaysian population. Whether OSA is higher or lower in patients with maxillary tori is not known.

ELIGIBILITY:
Inclusion Criteria:

* Complete edentulous patient with maxillary tori and without maxillary tori
* Complete edentulous patient who were willing give consent and eager to participate

Exclusion Criteria:

* Patients with swallow and mastication dysfunction
* Patients with cognitive disturbances
* Uncooperative patients.
* Patients with oral lesions, pathologies and Tempromandibular Joint disorders.
* Patients with systemic diseases
* Patients allergic to acrylic resin

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2018-09-17 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2020-09-16 (Actual)

PRIMARY OUTCOMES:
changes in the oral stereognosis | through study completion, an average of 1 year
  Oral stereognosis test will be performed using test pieces will be placed intraorally and patients will be instructed to identify the shape of test pieces with their tongue and palate. A visual representation chart of all 6 shaped forms will be provided to patient for identification purpose. Patients will be asked to identify the correct shape form by pointing out on the corresponding shape form on the chart. The 6 test pieces will be presented randomly to the patients and correct answer will not be informed to the patients during the OSA. The duration time for recognition of each shaped form for each patient will be noted and answers will be recorded on an OSA evaluation form. A correct answer will recorded as one point and incorrect answer is zero point. A full 6 points will be scored if all answers were correct. The response time and the OSA scores will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Indumathi Sivakumar, MDS, Principal Investigator — Senior Lecturer, Faculty of Dentistry, SEGi University, Malaysia
Locations (1):
- Faculty of Dentistry, SEGi University, Petaling Jaya, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: Yes
The data pertaining to oral stereognosis scores obtained by the participants and the response time duration for completing the test would be shared.
Supporting Information: Study Protocol
Time Frame: Data will be available from February 2020
Access Criteria: Researchers in this field of study who request data for multicentric study comparison. Data access request will be reviewed by a panel of reviewers.

REFERENCES:
- [Background] Ikebe K, Amemiya M, Morii K, Matsuda K, Furuya-Yoshinaka M, Nokubi T. Comparison of oral stereognosis in relation to age and the use of complete dentures. J Oral Rehabil. 2007 May;34(5):345-50. doi: 10.1111/j.1365-2842.2007.01687.x. PMID 17441875
- [Result] Park JH. Changes in oral stereognosis of healthy adults by age. J Oral Sci. 2017;59(1):71-76. doi: 10.2334/josnusd.16-0366. PMID 28367901
- [Result] Mantecchini G, Bassi F, Pera P, Preti G. Oral stereognosis in edentulous subjects rehabilitated with complete removable dentures. J Oral Rehabil. 1998 Mar;25(3):185-9. doi: 10.1046/j.1365-2842.1998.00221.x. PMID 9578225

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-09-17): https://cdn.clinicaltrials.gov/large-docs/48/NCT04254848/Prot_SAP_ICF_000.pdf